CLINICAL TRIAL: NCT04732208
Title: Validation of an Artificial Intelligence Model for Diabetic Retinopathy Screening Using a Smartphone-based Fundus Camera in the UK Population
Brief Title: Automated Screening of Diabetic Retinopathy Using a Smartphone-based Camera
Status: Completed | Type: Observational
Sponsor: Tameside General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: tgh001
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Retinopathy
Keywords: artificial intelligence; screening; fundus camera
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients
  Interventions: Diagnostic Test: Colour fundus photography

INTERVENTIONS:
Diagnostic Test: Colour fundus photography — Fundus images will be captured before and after administration of mydriatic agent
  Other Names: Instillation of mydriatic eye drops

SUMMARY:
The prevalence of diabetic retinopathy (DR) in the UK is on the rise. Within 20 years of diabetes diagnosis, nearly all people with type 1 and almost two thirds of people with type 2 diabetes (60%) have some degree of DR. NHS guidelines mandate annual DR screening in all patients aged 12 and above to prevent complications of DR. Screening for DR in England involves labour-intensive manual grading of retinal images through the teleophthalmology platform. Automated retinal image analysis systems with the use of artificial intelligence (AI) may offer an alternative to manual grading.

The purpose of this study is to evaluate the performance of a portable, hand-held fundus camera with integrated artificial intelligence for diabetic retinopathy screening by comparing it against the current standard i.e diagnosis provided by trained human graders evaluating the standard photographs/ophthalmologists.

DETAILED DESCRIPTION:
Study will enroll diabetic patients (new and established) meeting the inclusion criteria and who would provide an informed consent to participate in the study. This would include subjects who visit the endocrinology clinic and had either their retina evaluated by a teleophthalmology consult or visited the ophthalmology clinic for an indirect ophthalmoscopic fundus evaluation in the past 3 months. Subjects whose fundus has been recently evaluated in the past 3 months will also be re-called to the endocrinology clinic to get a fundus image captured on the Remidio NM FOP-10 device. Images will be captured by an operator who will be provided training in using the device prior to the study.

Non-mydriatic fundus images are captured using a pre-defined imaging protocol. One disc centered and one macula centred 45 deg image is taken for each eye. The images are then submitted to an AI system for analysis that runs locally on the Remidio FOP. An initial image quality assessment is performed by the AI. If the image is of sufficient quality then the AI will give an output of either 'signs of DR detected' (that would include moderate NPDR, severe NPDR, PDR and/or DME present) or no signs of diabetic retinopathy detected (that would include no DR, mild DR, absence of DME). If the image is of insufficient quality, then the operator makes 2 more attempts using the same imaging protocol. The images that are output as insufficient quality will be noted. All subjects who have provided consent for dilation are then instilled with a single drop of 1% tropicamide solution. After 20 mins, mydriatic 2 field (one disc centered and one macula centered) fundus images are captured and submitted to the AI for analysis along the same lines of non-mydriatic imaging. If the image is of insufficient quality then the operator makes 2 more attempts using the same imaging protocol. The images that are output as insufficient quality will be noted.

De-identified patient data including age, gender, ethnicity and lens status (Cataract grade, pseudophakia, aphakia) along with the final diagnosis made by a certified grader/ophthalmologist during clinical examination/teleophthalmology are retrieved from the NHS database. This DR diagnosis will act as a reference standard against which the AI output will be compared.

Data entry of subjects will be performed by approved trained Site Personnel. The de-identified data is stored onto an electronic data capture system (EDC). Approved Site Personnel will have a user specific log-in name and password to access the electronic data capture (EDC) system in order to enter study data. The principal investigator will ensure that all aspects of the study are complied with. The study will be conducted in accordance with applicable regulatory requirements and established rules for Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years who can provide an informed consent
* Established cases of diabetes mellitus (DM) with or without established diabetic retinopathy
* Subjects who have been dilated for an ophthalmic evaluation previously

Exclusion Criteria:

* Patients with acute vision loss
* Participants contraindicated for fundus imaging if hypersensitive to light or underwent recent photodynamic therapy or is photosensitive
* Participants who have been treated for diabetic retinopathy (laser or intra-vitreal injections) in the past 3 months
* Participants known to have other known retinal pathologies
* Participants identified to be at risk of acute angle closure glaucoma from previous ophthalmic evaluation (anterior chamber depth, gonioscopy to look at angles and IOP)
* Participants with known allergy to 1% tropicamide solution
* Currently participating in another investigational eye study and/or actively receiving investigational product for DR or diabetic macula edema.
* Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status- glycemic control, blood pressure etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with established diabetes mellitus presenting to GPs clinic for routine clinical care
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the AI in detecting any grade of diabetic retinopathy in those with established diabetes mellitus (DM) | 4 months

SECONDARY OUTCOMES:
To assess the positive predictive value, negative predictive value of AI in detecting any grade of DR | 4 months
To assess the sensitivity to identify sight-threatening diabetic retinopathy (STDR defined as severe NPDR or more severe disease and/or the presence of DME ie grades U, M1, R2 or R3) | 4 months
To compare the diagnostic ability of the AI in mydriatic and non-mydriatic eyes | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Edward Jude, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No